CLINICAL TRIAL: NCT07163377
Title: Effect of Art Therapy on Cognitive and Hand Functions of Alzheimer's Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, Assistant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90.2025fbu
Record Dates: First submitted 2025-08-20; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Art therapy; Cognitive Function
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy Session (Experimental): The intervention group will receive art therapy sessions over 8 weeks, twice weekly, each lasting 60 minutes. The program includes mandala coloring (weeks 1-2), collage making (weeks 3-4), clay modeling (weeks 5-6), free drawing/painting (week 7), and a participant's choice activity (week 8).
  Interventions: Other: Experimental Group
- Control Group (No Intervention): Participants in the control group will not receive any intervention

INTERVENTIONS:
Other: Experimental Group — Participants in the intervention group will undergo art therapy sessions
  Arms: Art Therapy Session

SUMMARY:
This randomized controlled trial aims to investigate the effects of art therapy on cognitive functions and hand functions in individuals with Alzheimer's disease. Alzheimer's disease is a progressive neurodegenerative disorder characterized by decline in memory, executive functions, and daily living activities. In addition, fine motor skills and hand-eye coordination are significantly impaired, limiting independence in daily tasks.

Art therapy is a non-pharmacological, low-cost, and feasible intervention that involves creative activities such as mandala painting, collage, clay modeling, and drawing. It has been shown to support cognitive performance, emotional well-being, and motor coordination by stimulating neuroplasticity. However, evidence focusing specifically on its impact on hand function in Alzheimer's patients remains limited.

In this study, 50 participants aged 60 years and older with mild to moderate Alzheimer's disease will be randomly assigned to an intervention group or a control group. The intervention group will attend art therapy sessions twice a week for 8 weeks (60 minutes per session), while the control group will receive no intervention. Cognitive functions will be assessed using the Mini-Mental State Examination (MMSE), and hand functions will be evaluated with the Nine Hole Peg Test (NHPT) and surface electromyography (sEMG) of forearm muscles.

The results of this study are expected to provide valuable evidence on the role of art therapy in supporting both cognitive and motor rehabilitation in Alzheimer's disease, potentially contributing to improved daily living independence and quality of life.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive neurodegenerative disorder characterized by impairments in memory, executive functions, attention, and activities of daily living. As the disease advances, fine motor skills and hand-eye coordination are also affected, limiting independence in self-care and functional tasks. Non-pharmacological approaches that target both cognitive and motor abilities are increasingly emphasized as complementary strategies to pharmacological treatment.

Art therapy is a creative intervention that incorporates activities such as mandala coloring, collage making, clay modeling, and drawing. Previous studies have shown that art therapy may stimulate neuroplasticity, improve attention and memory, reduce anxiety and behavioral symptoms, and enhance quality of life in individuals with dementia. However, limited evidence exists regarding its specific effects on fine motor performance and hand function in patients with Alzheimer's disease.

This randomized controlled trial is designed to evaluate the effectiveness of an 8-week structured art therapy program on cognitive functions and hand dexterity in individuals with mild to moderate Alzheimer's disease. Participants (n=50) will be randomly assigned to either an intervention group receiving art therapy twice weekly for 60 minutes per session, or a control group receiving no intervention.

Outcome measures include the Mini-Mental State Examination (MMSE) for global cognitive function, surface electromyography (sEMG) of forearm muscles to assess motor activity, and the Nine-Hole Peg Test (NHPT) to evaluate fine motor dexterity. Assessments will be conducted at baseline and post-intervention.

The study hypothesizes that participants in the art therapy group will demonstrate significant improvements in cognitive performance and fine motor abilities compared to the control group. The results are expected to provide evidence supporting the integration of art therapy as a feasible, low-cost, and non-pharmacological intervention in the rehabilitation of individuals with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years of age or older
* Having a diagnosis of mild or moderate Alzheimer's disease
* Possessing the physical and cognitive capacity to participate in art therapy interventions
* Providing informed consent

Exclusion Criteria:

* Being in the severe stage of Alzheimer's disease
* Having a history of severe psychiatric disorders such as schizophrenia or major depression
* Having a physical disability that prevents the use of the upper extremities
* Being unable to participate in the intervention due to visual or hearing impairments

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | From enrollment to the end of treatment at 8 weeks
  The Mini-Mental State Examination (MMSE) is a standardized test developed to assess the overall level of cognitive functioning in individuals. It is brief and easy to administer. The test consists of 11 items covering various cognitive domains, including orientation to time and place, short-term memory, attention and calculation, recall, language skills, and visuospatial abilities. The total score is 30; lower scores indicate cognitive impairment. In general, scores of 24 or below suggest the need for clinical attention regarding cognitive dysfunction.
Surface Electromyography (sEMG) | From enrollment to the end of treatment at 8 weeks
  The Mini-Mental State Examination (MMSE) is a brief, standardized instrument designed to evaluate global cognitive functioning in individuals. It can be administered in a short period of time and assesses 11 domains, including orientation to time and place, short-term memory, attention and calculation, recall, language abilities, and visuospatial skills. The maximum score is 30, with lower scores reflecting greater levels of cognitive impairment. A threshold score of 24 or below is generally considered indicative of clinically significant cognitive dysfunction warranting further evaluation.

SECONDARY OUTCOMES:
Nine Hole Peg Test | From enrollment to the end of treatment at 8 weeks
  The Nine-Hole Peg Test (NHPT) is a widely used, valid, and reliable performance test for assessing fine motor skills of the upper extremities. In the test, the participant is asked to place nine small pegs into a board with nine holes in a specific arrangement and then remove them one by one. The time taken to complete this task is measured with a stopwatch, and performance is evaluated based on this duration.

CONTACTS AND LOCATIONS:
Overall Officials: Mine SEYYAH, Ph.D., Principal Investigator — Fenerbahce University
Locations (1):
- Fenerbahçe Üniversitesi, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT07163377/Prot_SAP_000.pdf